CLINICAL TRIAL: NCT01537094
Title: The Effect of Vitamin C on Growth Hormone Secretion
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain funding to initiate the study. No subjects were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hideo Makimura, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-P-002912
Record Dates: First submitted 2012-02-10; First posted 2012-02-23 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Obese; Disorder of Vitamin C; Growth Hormone Secretion Abnormality
Keywords: low vitamin c; reduced growth hormone secretion
MeSH Terms: conditions — Obesity | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin C low dose (Active Comparator): vitamin C 250 mg oral once daily
  Interventions: Dietary Supplement: Vitamin C 250 mg once daily
- Vitamin C high dose (Active Comparator): vitamin C 1,000 mg oral once daily
  Interventions: Dietary Supplement: Vitamin C 1,000 mg once daily
- Placebo (Placebo Comparator): Placebo oral once daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Vitamin C 250 mg once daily
  Arms: Vitamin C low dose
Dietary Supplement: Vitamin C 1,000 mg once daily
  Arms: Vitamin C high dose

SUMMARY:
Obesity is associated with reduced growth hormone (GH) secretion. GH secretion is regulated by nutritional stimuli including fasting, insulin, glucose and free fatty acids. However, the role of micronutrients, such as vitamins, on GH secretion has not been investigated in much detail. Vitamin C levels are also reduced in obesity, and the investigators recently demonstrated a possible role for dietary vitamin C intake in the regulation of GH secretion in two preliminary retrospective studies. The investigators therefore propose a more detailed prospective physiological study to examine the effects of increasing dietary vitamin C intake on GH secretion in a physiologic, intervention study. The investigators hypothesize that increasing vitamin C concentrations in obese subjects with sub-optimal plasma vitamin C levels and reduced GH secretion will increase GH secretion.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-60
2. BMI ≥ 30 kg/m2
3. Waist circumference ≥ 102 cm in men and ≥ 88 cm in women
4. Plasma vitamin C concentration ≤ 23 µmol/l
5. Peak stimulated GH ≤ 4.2 µg/l upon GHRH-arginine stimulation test

Exclusion Criteria:

1. History of hypopituitarism, pituitary surgery, pituitary/brain radiation, recent traumatic brain injury or any other condition known to affect the GH axis.
2. History of severe chronic illness including anemia, chronic kidney disease, liver disease, oxygen dependent COPD or HIV
3. Subjects on testosterone, glucocorticoids, anabolic steroids, GHRH, GH or IGF-1 within 3 months of enrollment
4. Use of dietary supplements including vitamin C or once daily multi-vitamins
5. Subjects with Hgb < 912 g/dL, SGOT > 2.5x upper limit of normal or Creatinine > 1.5 mg/dL
6. Subjects with poorly controlled diabetes, defined as HbA1c > 8%.
7. Changes in lipid lowering or anti-hypertensive regimen within 3months of screening
8. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit
9. Any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in GH secretion at 4 weeks | Change from Baseline to 4 weeks
  GH secretion will be assessed by overnight frequent blood sampling to assess maximum GH, nadir GH, mean overnight GH, as well as parameters of pulsatile secretion.

CONTACTS AND LOCATIONS:
Overall Officials: Hideo Makimura, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States